CLINICAL TRIAL: NCT05781607
Title: A Retrospective Cohort Study on the Long-term Efficacy and Influencing Factors of Physical Therapy for Temporomandibular Joint Disorders
Brief Title: Long-term Efficacy of Physical Therapy for TMDs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: SH9H-2022-T162-2
Record Dates: First submitted 2023-03-12; First posted 2023-03-23 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-03

CONDITIONS: Temporomandibular Joint Disorders
Keywords: temporomandibular joint disorders; physical therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PE: Patient education combined with drug therapy group
  Interventions: Combination Product: Patient education combined with drug therapy
- PT: Individualized comprehensive physical therapy group
  Interventions: Combination Product: Individualized comprehensive physical therapy

INTERVENTIONS:
Combination Product: Patient education combined with drug therapy — Receive a health education by a specialist therapist, including explaining the anatomy and function of TMJ; Explain the etiology, prognosis, treatment plan and prognosis of TMD; Correct the patients' daily oral habits, such as unilateral chewing, habitual clenching, eating too much hard food, etc; Instruct the patient to understand the rest position of the temporomandibular joint and correct the bad posture of the neck and shoulder. At the same time, corresponding medication should be given, and NSAIDS should be taken orally or externally for patients with pain.
  Groups: PE
Combination Product: Individualized comprehensive physical therapy — Physical factor therapy and/or manual therapy
  Groups: PT

SUMMARY:
Physical therapy is one of the initial conservative treatments for TMD. Many studies and previous studies in our department have proved that it can improve the pain, mouth opening and mandibular function of patients with TMD. However, the current research on physical therapy for TMD has a short follow-up period, which cannot prove that the patients' long-term mandibular function has improved, and few studies have analyzed the relevant factors affecting the curative effect. Therefore, this study is intended to adopt a retrospective cohort study to include TMD patients who received physical therapy in our department from 2016.01-2021.12. The patients' pain, joint area noise, mandibular range of motion, mandibular function and other conditions will be followed up by remote telephone or online questionnaire, and the patients' demography, clinical symptoms, pain, oral habits, depression, anxiety, sleep status, head and neck posture and other information will be collected. The multiple regression analysis model will be used to compare and analyze the relevant factors affecting the prognosis of patients, and to intervene in advance the factors that have a significant impact on the prognosis of the disease, so as to improve the treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* The first-episode TMD patients with pain, limited mouth opening and abnormal noise in the joint area; 12-80 years old; regardless of gender; The patient received physical therapy in the outpatient department; MRI or CBCT imaging was completed before enrollment

Exclusion Criteria:

* Patients with recurrent TMD; Patients who had previously undergone TMJ surgery; Patients with nervous system diseases, immune system diseases, tumors and other diseases that the attending physician considers unsuitable for inclusion in the study; Cognitive impairment

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: TMD patients who received patient education or physical therapy in the Department of Rehabilitation Medicine of the Ninth People's Hospital affiliated to Shanghai Jiaotong University Medical College from January to December 2016
Sampling Method: Probability Sample
Enrollment: 189 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2024-04-06 (Estimated); Study Completion 2024-06-06 (Estimated)

PRIMARY OUTCOMES:
Long term effective rate | 12 months
  Long-term effective rate=number of effective cases/total number of cases

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
After the research results are published, the original data will be shared in the form of network data sets

REFERENCES:
- [Derived] Jin L, Yao Y, Fang Z, Fan S, Cai B, Xu L, Liu S. Long-Term Prognosis and Influencing Factors of Chinese Adolescents With Temporomandibular Disorder After Physical Therapy. J Oral Rehabil. 2024 Dec;51(12):2611-2621. doi: 10.1111/joor.13865. Epub 2024 Sep 20. PMID 39305035